CLINICAL TRIAL: NCT07063069
Title: Evaluation of the Value of Ultrasound Measurement of Stomach Diameter in Predicting Postoperative Nausea/Vomiting
Acronym: EVOL2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 49RC24_0252; 2025-A00733-46 (Other: ANSM)
Record Dates: First submitted 2025-06-12; First posted 2025-07-14 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Patient With Indication for Major Abdominal Submesocolic, Parietal, Left Pancreatic or Liver Surger

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Abdominal ultrasound (Experimental): All patients included will have an abdominal ultrasound scan
  Interventions: Other: Abdominal ultrasound

INTERVENTIONS:
Other: Abdominal ultrasound — All patients included will have an abdominal ultrasound scan to mesure anterior/posterior external diameter of gastric antrum upstream of pyloru and external diameter upper/lower of gastric antrum upstream of pylorus

SUMMARY:
The advent of enhanced rehabilitation after surgery has helped to reduce surgical stress, thereby improving postoperative outcomes by reducing the time it takes for patients to recover their transit and autonomy.

Despite this, some 10-30% of patients undergoing abdominal surgery will experience postoperative ileus or nausea/vomiting. In addition to increasing the length of hospital stay, these complications increase patient discomfort and, above all, the risk of inhalation pneumonitis.

With the advent of enhanced rehabilitation, patients are receiving less drainage, particularly nasogastric drainage, which is now virtually outlawed in scheduled sub-mesocolic abdominal surgery.

In a recent international multicenter study of patients undergoing colorectal surgery, the authors reported that less than 10% of patients received a nasogastric tube routinely, and that 20% received it for clinical reasons (before or after nausea/vomiting). The authors also reported an overall inhalation pneumonitis rate of 4.2%. The authors concluded from this study that nasogastric tubes should not be inserted routinely, but that delay in nasogastric tube insertion was a risk factor for pneumopathy.

As the onset of postoperative pneumopathy is associated with a risk of mortality, it seems important to predict its risk of onset in order to target patients who could benefit from early nasogastric tube placement.

A recent study carried out in the visceral surgery department of the CHU d'Angers evaluated the evolution of gastric distension. One of the objectives of the ancillary study was to evaluate the interest of the ratio of gastric antrum distension measurement in 2 axes (longitudinal and axial) at D2 postoperative / D preoperative.

As this was an ancillary study of a preliminary study, the number of events was 12, making it impossible to assert with high power that the appearance of nausea/vomiting is linked to the ratio described above. An observational study including more patients is therefore needed to confirm this hypothesis before carrying out a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* Indication for major abdominal surgery (submesocolic, parietal, left pancreas or liver)
* Patient affiliated to or benefiting from a social security scheme

Non-inclusion criteria

* Patient refusal to participate in study
* Need for immediate post-operative ICU stay
* Surgery performed as an emergency
* Esophageal, gastric or cephalic pancreatic surgery
* Person deprived of liberty by judicial or administrative decision
* Person under compulsory psychiatric care

Exclusion Criteria:

* Discharge with nasogastric tube
* Immediate admission to post-operative intensive care unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Evaluate the sensitivity and specificity of the diagnostic character of the gastric diameter ratio at Day 2 / Day 0 | Day 2/Day 0 after surgical intervention
  Postoperative ileus is defined according to the Vather et al. criteria.

SECONDARY OUTCOMES:
assess the sensitivity and specificity of the gastric diameter ratio at D2/D0 in predicting the onset of inhalation pneumonitis | Day 2/Day 0 after surgical intervention
  the onset of inhalation pneumonitis, defined as a cough with varying degrees of fever secondary to surgery. Inhalation pneumonitis is clinically suspected and confirmed on imaging with a standard chest X-ray
code a computer program to automatically measure the diameter of the gastric antrum | Day 2/Day 0 after surgical intervention
  Gastric antrum diameter measurements and images

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Angers, Angers, France

IPD SHARING:
Plan to Share IPD: No